CLINICAL TRIAL: NCT04499287
Title: Mealtime Walking Study to Improve Postprandial Metabolic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OxPMW
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: PreDiabetes; Postprandial Hyperglycemia
Keywords: blood glucose; blood insulin; fiber; prediabetes; postprandial glycemia
MeSH Terms: conditions — Prediabetic State; Hyperglycemia | interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: randomized, controlled, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Test meal [bagel with butter (20 g) and apple juice (240 ml) with added sugar (24 g)] The meal was a total of 640 kcal (100 g carbohydrate, 21 g fat, 10 g protein. Participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption. One week later the test meal was consumed with fiber (36 g, Metamucil powder, Procter&Gamble, Cincinnati, OH) added to the apple juice (active) and participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption . One week later participants were given 5 minutes to transition to the treadmill following consumption of the test meal and began walking on a motorized treadmill at their calculated preferred walking speed for 15 minutes (experimental). Afterwards participants remained seated in the laboratory with minimal activity for the remainder of the four hours following test meal consumption
  Interventions: Other: 15-minute walk at preferred walking speed.; Dietary Supplement: Fiber; Other: control
- Fiber (Active Comparator): Test meal [bagel with butter (20 g) and apple juice (240 ml) with added sugar (24 g)] The meal was a total of 640 kcal (100 g carbohydrate, 21 g fat, 10 g protein. 9 grams of soluble viscous fiber from psyllium husk (36 g, Metamucil powder, Procter&Gamble, Cincinnati, OH) was mixed with the apple juice. Participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption. One week later participants were given 5 minutes to transition to the treadmill following consumption of the test meal and began walking on a motorized treadmill at their calculated preferred walking speed for 15 minutes (experimental). Afterwards participants remained seated in the laboratory with minimal activity for the remainder of the four hours following test meal consumption. One week later the test meal was consumed, and participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption (placebo).
  Interventions: Other: 15-minute walk at preferred walking speed.; Dietary Supplement: Fiber; Other: control
- Walk (Experimental): Test meal [bagel with butter (20 g) and apple juice (240 ml) with added sugar (24 g)] The meal was a total of 640 kcal (100 g carbohydrate, 21 g fat, 10 g protein. Participants were given 5 minutes to transition to the treadmill following consumption of the test meal and began walking on a motorized treadmill at their calculated preferred walking speed for 15 minutes. Afterwards participants remained seated in the laboratory with minimal activity for the remainder of the four hours following test meal consumption One week later the test meal was consumed, and participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption (placebo comparator). One week later the test meal was consumed with fiber (36 g, Metamucil powder, Procter&Gamble, Cincinnati, OH) added to the apple juice and participants remained seated in the laboratory with minimal activity for the four hours following test meal consumption (active comparator).
  Interventions: Other: 15-minute walk at preferred walking speed.; Dietary Supplement: Fiber; Other: control

INTERVENTIONS:
Other: 15-minute walk at preferred walking speed.
Dietary Supplement: Fiber — 9 grams soluble fiber
Other: control — control

SUMMARY:
This randomized crossover trial will investigate the metabolic responses following the consumption of a bagel+juice meal under 3 conditions: control, fiber (positive control), and postmeal walk in15 healthy adults. It is hypothesized that the postmeal walk will reduce glycemia, insulinemia, and oxidative stress similar to fiber.

DETAILED DESCRIPTION:
The study will follow a randomized, crossover design. Participants and the investigator will be blinded for the control treatments but not for the walk treatment. Participants will complete 3 meal tests; tests are separated by about 1 week. An initial screening visit will be scheduled for the online survey respondents that meet the inclusion criteria and are willing to consider participation. At this visit, written consent will be secured followed by further screening for the exclusion criteria and the collection of demographic and health history data and anthropometric measures. A fasting blood sample will be collected for glucose analysis. Participants will be scheduled for experimental testing and provided with instructions and calendars. Participants will be given at least one week's notice if they do not qualify for the trial based on fasting glucose concentrations.

On the day prior to each experimental day, the participants will consume 2 bagels (54 g carbohydrate/bagel), and on the night prior to each visit, participants will consume a standard dinner of their choice. (The bagels will be provided to participants and the standardized dinner will be documented. The bagels and standardized dinner meal will facilitate controlled 'glycogen loading' prior to testing.) No other food will be consumed after this dinner meal, and participants will fast overnight until they arrive at the research center the next morning (e.g., no food or beverage with the exception of water). Fasting blood (1 tablespoon) will be collected and the test meal (bagel+juice) will be consumed. Postprandial blood samples will be collected for 4 hours (see below). The subjects will not be allowed to consume any food or beverage (with the exception of water) through the duration the visit. A snack will be provided to participants once the testing is over.

Glucose: 0,15,30,60,120, 180, 240 Insulin: 0, 30, 120, 180, 240 Oxidative Stress Markers: 0, 180, 240

The blood insulin level will be determined in venous blood by RIA. Capillary blood glucose will be determined with a glucometer. Oxidative stress, e.g., total antioxidant capacity, IL-6, and TBARS will be assessed using microplate analyses kits.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI ≥ 30 kg/m2)
* nonsmoking
* sedentary
* fasting capillary blood glucose that measured from 5.6 to 6.9 mmol/L

Exclusion Criteria:

* answered "yes" to any of the questions on the "Par-Q & You" questionnaire
* refused to discontinue antioxidant supplement use for several weeks prior to and during the study
* prescribed medication use (unless use was consistent for the 3 months prior to the study and intake remained consistent throughout the study duration)
* food allergies or medical conditions that impacted normal functioning of the gastrointestinal tract

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2015-02-14 (Actual); Study Completion 2015-03-10 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | 4 hours
  incremental area under curve
postprandial insulinemia | 4 hours
  incremental area under curve

SECONDARY OUTCOMES:
postprandial oxidative stress | 4 hours
  total antioxidant capacity of blood
postprandial oxidative stress | 4 hours
  blood interleukin-6
postprandial oxidative stress | 4 hours
  Thiobarbituric Acid Reactive Substances TBARS

IPD SHARING:
Plan to Share IPD: No